CLINICAL TRIAL: NCT00300716
Title: Double Blind Placebo Controlled Pilot Trial of Memantine for Cognitive Impairment in Multiple Sclerosis
Brief Title: Trial of Memantine for Cognitive Impairment in Multiple Sclerosis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: Forest Laboratories (Industry); University of Southern California (Other); University of Texas Southwestern Medical Center (Other); MS-Hub Seattle (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NAM-MD-13
Record Dates: First submitted 2006-03-08; First posted 2006-03-09 (Estimated); Last update posted 2019-10-15 (Actual); Status verified 2019-10

CONDITIONS: Multiple Sclerosis; Cognition Disorders
Keywords: Multiple Sclerosis; Cognitive impairment; Memantine; Placebo; Neuropsychological tests; Quality of life; Fatigue
MeSH Terms: conditions — Multiple Sclerosis; Cognition Disorders; Cognitive Dysfunction; Fatigue | interventions — Memantine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Memantine

SUMMARY:
This study is designed to determine whether memantine is an effective treatment for memory and cognitive problems associated with multiple sclerosis when compared to placebo.

DETAILED DESCRIPTION:
Objective:

The objective of this pilot project is to conduct a clinical trial to assess the efficacy of memantine as a treatment for cognitive dysfunction in multiple sclerosis (MS). We hypothesize that MS patients with cognitive impairment treated with memantine will demonstrate an improvement in performance on a neuropsychological test battery as compared to placebo treated patients.

Background and Significance:

Cognitive dysfunction is a major cause of disability in multiple sclerosis (MS). The estimated prevalence of cognitive dysfunction in the MS population is 45% to 65%. MS patients with cognitive dysfunction have fewer social interactions, more sexual dysfunction, greater difficulty with household tasks and higher unemployment than those with normal cognition. At present, there is no effective pharmacological symptomatic treatment for the cognitive dysfunction of MS. One agent that may have some benefit in treating this condition is the N-methyl-D-aspartate (NMDA) receptor antagonist memantine.

Memantine is a NMDA antagonist that has been shown to be effective in treating Alzheimer's disease. Glutamate toxicity has been implicated in the pathogenesis of a variety of neurologic diseases, including MS. Glutamate receptor activation may be involved both in mediation of neural injury and in neuronal dysfunction. By blocking NMDA receptors, memantine may both improve neuronal function, explaining symptomatic improvement in some Alzheimer's patients, and slow progressive neuronal death, potentially resulting in a slowing of cognitive decline in Alzheimer's patients. The pathogenesis of cognitive dysfunction in MS relates at least in part to the extent of cerebral demyelination, axonal loss and atrophy. Some cognitive dysfunction is reversible. Reduction in inflammation can result in improvement in cognitive performance. What role NMDA receptors and glutamate toxicity may play in cognitive dysfunction is uncertain but, given the lack of any treatment for cognitive dysfunction in MS, performing a pilot trial of memantine in MS is clearly warranted.

Overall Design:

This is a placebo-controlled, double-blinded, randomized, parallel-group pilot study of 16 weeks duration in MS patients with cognitive impairment. There will be 73 patients per treatment arm among all sites. The intervention arm will receive 20 mg of memantine a day. Randomization into each treatment arm will be stratified on age and CVLT score. A double-blind, placebo controlled trial is critical to perform even for a pilot trial. Both learning and placebo effect are likely to improve the cognitive performance of some subjects. An open labeled trial would likely show some improvement in the patients but the results would not be interpretable.

Memantine:

Both memantine and the placebo will be provided by Forest Laboratories Inc.

Scheduled Visits:

Visit 1:

The subject will receive a consent form. After signing, visual acuity will be tested. The Multiple Sclerosis Screening Neuropsychological Questionnaire (MSNQ) and the Modified Neuropsychiatric Inventory (MNPI) will be given to the primary caregiver if present, or to the patient instructing him to have the primary caregiver fill it out and return it in the next visit. They will receive the first half of the neuropsychological test battery, which includes the Paced Auditory Serial Addition Test (PASAT) and California Verbal Learning Test II (CVLT-II). They will also receive the Beck Depression Inventory (BDI). Women of childbearing potential will be asked to give a urine sample for a pregnancy test (beta HCG). At this point, patients will be informed whether they have met the full criteria for enrollment. If they qualify then they will receive the second half of the neuropsychological tests (Controlled Oral Word Association Test, Stroop Color And Word Association Test, Symbol Digit Modalities Test and Delis-Kaplan Executive Function System). This visit will last approximately 1½ hour if the patient does not qualify for the study and 2 hours if they qualify.

Visit 2:

The subjects will receive the Fatigue Severity Scale (FSS), Modified Fatigue Impact Scale (MFIS), the Medical Outcomes Study 36 Item Short Form Health Survey (SF-36) and the Perceived Deficits Questionnaire (PDQ) from the Multiple Sclerosis Quality of Life Inventory (MSQLI). A physical exam and a neurological exam will be performed. Memantine and placebo pills will be dispensed; the neurological exam will include the Expanded Disability Status Scale, a 25 feet timed walk and the nine-hole peg test. The starting dose of memantine will be 5 mg once daily. The dose will be increased in 5 mg increments to 10 mg/day (5 mg twice a day), 15 mg/day (5 mg and 10 mg as separate doses), and 20 mg/day (10 mg twice a day) over 4 weeks and then continued at 20 mg for the rest of the study. In case of intolerable side effects when titrating the dose up the dose can be decreased to the previously tolerated dose. This visit will last 1 1/2 hours.

Telephone follow-up:

Four telephone follow-up visits will be carried-out for all enrolled subjects between Visits 2 and 3. These will occur at two weeks after Visit 2 and again at four, seven, and eleven weeks after Visit 2. These calls will review study procedures, check for compliance and reports of side effects. The person calling should be different from the person that administers the neuropsychological tests. The total time for the telephone visit is 15 minutes.

Side effect evaluation visit:

If any unexpected side effects occur, subjects will be evaluated with a physical exam and a neurological exam. This visit will last approximately 1 hour. Relapses will be documented as adverse events and the evaluation will include the EDSS, timed walk and 9 hole peg test.

Visit 3:

Subjects will return to clinic for the final assessment 4 weeks after the last telephone follow-up visit. At this visit, subjects will complete the full neuropsychological test battery. The SF-36 and PDQ, BDI, FSS, and MFIS will be administered. The MSNQ and the MNPI will be given to the caregiver. A repeat neurological and physical exam will be performed. This visit will last 2 ½ hours.

ELIGIBILITY:
Inclusion Criteria:

1. A diagnosis of multiple sclerosis as defined by the McDonald criteria. Patients with relapsing-remitting, secondary progressive, and primary progressive forms of MS are eligible.
2. Age between 18 and 65 years.
3. Demonstrated cognitive dysfunction at screening defined as a score worse than 1.0 standard deviations below the mean on the PASAT or the CVLT-II.

Exclusion Criteria:

1. A history of major depression, psychosis, or a score > 19 on the Beck's Depression Inventory.
2. Corrected binocular visual acuity worse than 20/50; any impairment of binocular color vision.
3. Patients that do not speak English as a primary language (fluency may impact performance).
4. A clinically significant MS exacerbation within 30 days of the screening
5. Pregnancy
6. Renal insufficiency.
7. History of seizures.
8. Patients using acetazolamide (Diamox, Ak-sol, Storzolamide), dichlorphenamide (Daranide), methazolamide (Neptazane) or topiramate (Topamax), dextromethorphan (Robitussin DM and other cold remedies), or amantadine (Symmetrel).
9. Use of medical marijuana in the prior six months.
10. History of alcohol abuse or illicit drug use in the prior six months.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2004-04; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Change in the Paced Auditory Serial Addition Test and the California Verbal Learning Test II (multivariate end-point) after 15 weeks of treatment.

SECONDARY OUTCOMES:
Controlled Oral Word Association Test
Stroop Color and Word Test
Symbol Digit Modalities Test
Delis-Kaplan Executive Function System
Perceived Deficit Questionnaire
Multiple Sclerosis Screening Neuropsychological Questionnaire
Modified Neuropsychiatric Inventory
Fatigue Severity Scale
Modified Fatigue Impact Scale
MS Quality of Life Inventory
Beck Depression Inventory

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Bourdette, MD, Principal Investigator — Oregon Health and Science University; Lovera Jesus, MD, Principal Investigator — Oregon Health and Science University; Daniel Bandari, MD, Principal Investigator — University of Southern California; Ted Brown, MD, Principal Investigator — MS Hub; Elliot Frohman, MD, Principal Investigator — UT Southwestern
Locations (4):
- United States (4):
  - USC, Los Angeles, California
  - OHSU, Portland, Oregon
  - UT Southwestern, Dallas, Texas
  - MS Hub, Seattle, Washington

REFERENCES:
- [Derived] Lovera JF, Frohman E, Brown TR, Bandari D, Nguyen L, Yadav V, Stuve O, Karman J, Bogardus K, Heimburger G, Cua L, Remingon G, Fowler J, Monahan T, Kilcup S, Courtney Y, McAleenan J, Butler K, Wild K, Whitham R, Bourdette D. Memantine for cognitive impairment in multiple sclerosis: a randomized placebo-controlled trial. Mult Scler. 2010 Jun;16(6):715-23. doi: 10.1177/1352458510367662. Epub 2010 May 18. PMID 20483885
- See also: Related Info — http://www.ohsu.edu/xd/health/clinical-trials/clinical-trial-results.cfm